CLINICAL TRIAL: NCT05365113
Title: Comparison of Hemodynamic Effects of Two Modalities of Alveolar Recruitment Maneuvers in Major Abdominal Surgery Patients: A Physiological Study
Brief Title: Comparison of Hemodynamic Effects of Two Modalities of Alveolar Recruitment Maneuvers in Major Abdominal Surgery Patients
Acronym: CHARM-Bloc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RBHP 2021 GODET 4 (Charm Bloc)
Record Dates: First submitted 2022-04-19; First posted 2022-05-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Output; Decreased Cardiac Output; Hemodynamic Monitoring; Blood Pressure; Stroke Volume; Major Abdominal Surgery; Mechanical Ventilation; Hemodynamic Optimization
Keywords: mechanical ventilation,; hemodynamics,; ARM,; CPAP,; extended sigh,; cardiac output
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Intervention Model Description: Exploratory study testing in cross-sectional design two alveolar recruitment maneuvers referenced in practice, in patients under general anesthesia and intubated under controlled ventilation, in operating room
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous positive airway pressure (CPAP) then extended sigh (Active Comparator): Patients assigned to this group will receive a CPAP ARM (40cmH2O during 50 seconds), followed by a 10-minute pause corresponding to a period of return to basal state.
  Then an ARM by extended sigh (e-sigh) also 50 seconds (driving pressure at 10cmH2O and successive PEEP levels at 10, 15, 20, 25 and 30cmH2O, with respiratory frequency fixed at 30/min in controlled pressure).
  Hemodynamic (blood pressure, cardiac output, stroke volume) and ventilatory measurements will be performed the last 10 seconds of each recruitment maneuver.
  Interventions: Procedure: alveolar recruitment maneuver
- extended sigh then continuous positive airway pressure (CPAP) (Active Comparator): Patients assigned to this group will receive an ARM by extended sigh (e-sigh) during 50 seconds (driving pressure at 10cmH2O and successive PEEP levels at 10, 15, 20, 25 and 30cmH2O, with respiratory frequency fixed at 30/min in controlled pressure), followed by a 10-minute pause corresponding to a period of return to basal state.
  Then they receive a CPAP ARM (40cmH2O during 50 seconds). Hemodynamic (blood pressure, cardiac output, stroke volume) and ventilatory measurements will be performed the last 10 seconds of each recruitment maneuver.
  Interventions: Procedure: alveolar recruitment maneuver

INTERVENTIONS:
Procedure: alveolar recruitment maneuver — When patient is under general anesthesia, an arterial catheter is placed for cardiac output and stroke volume (SV) monitoring. To avoid pre-load dependency bias, the blood volume will be optimized. A 250mL fluid-challenge of a balanced crystalloid solution is administered under cover of the SV monitoring. If SV variation is greater than 10%, a new fluid-challenge is performed to obtain a reference SV, corresponding to the patient's optimal blood volume.The patient is then "pre-load independent".
  Then, patients will be randomized into two groups: a first group will receive a CPAP ARM: 40 cmH2O for 50 seconds, followed by a 10-minute break corresponding to a period of return to basal state; then an extended sigh ARM (e-sigh) also lasting 50seconds (driving pressure: 10cmH2O and successive PEEP levels at 10,15,20,25 and 30cmH2O, a respiratory rate set at 30/min in controlled pressure - 5cycles at each PEEP level); a second group will receive the same two ARM modalities in reverse order.

SUMMARY:
The objective of this study is to investigate the hemodynamic effects of two strategies of alveolar recruitment maneuver in patients undergoing major abdominal surgery in the operating room

DETAILED DESCRIPTION:
In practice, after induction of general anesthesia and intubation, patients will be conditioned with the recommended monitoring (arterial catheter, central venous catheter, and transpulmonary thermodilution).

Once conditioning is complete, optimization of blood volume will be performed with volumetric expansions (250 mL of Ringer lactate) to achieve a change in stroke volume of less than 10%, as recommended (RFE SFAR 2013 - Perioperative Vascular Filling Strategy). The patient will then be randomized to one of the following groups: [ extended sigh then CPAP ] or [ CPAP then extended sigh ] (random order of ARMs - each patient becoming their own control). In order to homogenize the settings, the mechanical ventilation will be standardized with in particular the use of a PEEP of 6 cmH2O before inclusion and between the ARMs (for a duration of at least 10 minutes in each case).

Hemodynamic values will be recorded during the last 10 seconds of each procedure. Once the two ARMs have been performed, the rest of the management will then be left to the discretion of the practitioner in charge of the patient.

The included patient will be managed according to the recommendations at the time of the study.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old
* patient under general anesthesia
* patient intubated under controlled invasive mechanical ventilation
* patient with invasive hemodynamic monitoring (transpulmonary thermodilution)
* patient sedated (BIS between 40 and 60) and/or curarized with TOF monitoring to avoid inspiratory effort
* patient optimized on the hemodynamic level, in particular with regard to blood volume, following the hemodynamic monitoring data and the recommendations of the French Society of Anesthesia and Resuscitation (RFE SFAR 2013 - Perioperative vascular filling strategy)
* patient covered by a Social Security plan
* patient consent to participate in the study

Exclusion Criteria:

* contraindication to the use of cardiac output measurement
* cardiac arrhythmia
* pace-maker/implantable defibrillator
* severe valvulopathy
* contraindication to the use of the tomographic electroimpedancemetry technique
* thoracic lesions, thoracic dressing
* left ventricular ejection fraction (LVEF) < 45% and/or right ventricular failure.
* history of pulmonary lobectomy and/or pneumonectomy and/or known emphysema
* patient with restrictive or obstructive lung disease
* body mass index (BMI) < 16.5 or > 30 kg.m-2
* pregnancy
* intracranial hypertension or suspected intracranial hypertension
* patient under limitation of care
* patient under legal protection (guardianship, curatorship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the change in cardiac output during the last 10 seconds of each MRA modality from its baseline value (determined after hemodynamic optimization and before the procedure was performed) | last 10 seconds of each ARM modality
  Cardiac output (l/min) will be measured by invasive monitoring during the last 10 seconds of each recruitment maneuver

SECONDARY OUTCOMES:
Standard hemodynamic monitoring data | last 10 seconds of each ARM modality
  blood pressure, mean arterial pressure,
Standard hemodynamic monitoring data | last 10 seconds of each ARM modality
  heart rate
Invasive hemodynamic monitoring data | last 10 seconds of each ARM modality
  stroke volume change in stroke volume
Invasive hemodynamic monitoring data | last 10 seconds of each ARM modality
  change in stroke volume
Evaluation of standard ventilatory monitoring data | last 10 seconds of each ARM modality
  tidal volume (ml)
Evaluation of standard ventilatory monitoring data | last 10 seconds of each ARM modality
  positive end-expiratory pressure (PEEP), peak pressure, plateau inspiration pressure, driving pressure
Evaluation of standard ventilatory monitoring data | last 10 seconds of each ARM modality
  respiratory rate,
Evaluation of standard ventilatory monitoring data | last 10 seconds of each ARM modality
  inspired oxygen fraction,
Evaluation of standard ventilatory monitoring data | last 10 seconds of each ARM modality
  compliance of the respiratory system
Electro-impedancemetry data | last 10 seconds of each ARM modality
  Analysis of pulmonary aeration will be performed using the non-invasive technique of tomographic electroimpedancemetry with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  COV : Center Of Ventilation and GI : Global Inhomogeneity index
Electro-impedancemetry data | last 10 seconds of each ARM modality
  Analysis of pulmonary aeration will be performed using the non-invasive technique of tomographic electroimpedancemetry with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  TIV : Tidal Impedance Variation
Electro-impedancemetry data | last 10 seconds of each ARM modality
  Analysis of pulmonary aeration will be performed using the non-invasive technique of tomographic electroimpedancemetry with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  RVD : Regional Ventilation Delay
Electro-impedancemetry data | last 10 seconds of each ARM modality
  Analysis of pulmonary aeration will be performed using the non-invasive technique of tomographic electroimpedancemetry with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  EELI : End Expiratory Lung Impedance
Electro-impedancemetry data | last 10 seconds of each ARM modality
  Analysis of pulmonary aeration will be performed using the non-invasive technique of tomographic electroimpedancemetry with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  percentages of overdistended and atelectasis areas
Paraclinics data | last 10 seconds of each ARM modality
  During the last 10 seconds of the recruitment maneuver, capnography will be recorded
Paraclinics data | last 10 seconds of each ARM modality
  During the last 10 seconds of the recruitment maneuver, SpO2 will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Clermont-Ferrand, France